CLINICAL TRIAL: NCT06510244
Title: Measuring Pain Perception to the Same Stimulus in Different Patients Using Electroencephalography and Numerical Rate Scale
Brief Title: Pain Perception Measurement by EEG and NRS
Status: Recruiting | Type: Observational
Sponsor: Cleveland Dental Institute (Other)
Responsible Party: Sponsor
Other Study IDs: CDIENDO0002
Record Dates: First submitted 2024-07-15; First posted 2024-07-19 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Pain; Electroencephalography; Toothache
Keywords: pain perception; Numeric Pain Rating Scale; electroencephalography
MeSH Terms: conditions — Pain; Toothache | interventions — Dental Pulp Test

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- One group of patients between 20-60 years old: Patients between 20-60 years old with a tooth health and no history of dental alveolar trauma or pulp chamber calcification.
  Interventions: Device: EEG EMOTIV

INTERVENTIONS:
Device: EEG EMOTIV — The teeth will be dried with 2x2 gauze; then, Endo Ice will be applied. The patient response will be written on a sheet numbering to choose from 0 to 10, and at the same time, the brain waves will be recorded through EEG.
  Other Names: Noninvasive Electroencephalography; Endo-Ice

SUMMARY:
Observational study at CDI Cleveland Dental Institute. Investigators will assess the pain perception in one group of patients using two non-invasive methods. First, a numerical rate scale (NRS) and second, a brain wave EEG.

DETAILED DESCRIPTION:
To generate the nociceptive stimulus, The investigators will apply cold (Endo-Ice) to a healthy upper incisor tooth #8. Inclusion criteria: Patients between 20 and 60 years old, with healthy teeth, no history of dental alveolar trauma, and no pulp chamber calcification. After the nociceptive stimulus, patients will write their pain perception on paper from 0 to 10, and at the same time, we will record the brain activity with a non-invasive EEG Emotiv. Then, we will correlate both methods.

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* Age: 20-60 years.
* Tooth #8 vital and mature. No history of dentoalveolar trauma.
* Adequate coronal tooth structure.

Exclusion Criteria:

* Chronic periodontitis.
* Vertical root fracture.
* Immature teeth.
* Necrotic teeth.
* Systemic diseases that affect the healing process.
* Non restorable teeth.

Ages: 20 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: In the outpatient clinic of CDI Cleveland Dental Institute, patients with mature and vital tooth #8 are between 20 and 60 years old.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Pain Perception Measurement by EEG. | January 2024-December 2024
  to observe the brain waves changes during pain perception
Pain Perception Measurement by EEG and NRS. | January 2024-December 2024
  To establish a possible correlation between the NRS and EEG measurements.

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Dental Institute, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alcock MM. Defining pain: past, present, and future. Pain. 2017 Apr;158(4):761-762. doi: 10.1097/j.pain.0000000000000828. No abstract available. PMID 28301403
- [Background] Matsuda S, Itoi H, Ryoke T, Yoshimura H. How should clinicians assess acute dental pain?: A review. Medicine (Baltimore). 2022 Nov 11;101(45):e31727. doi: 10.1097/MD.0000000000031727. PMID 36397373
- [Background] Mouraux A, Iannetti GD. The search for pain biomarkers in the human brain. Brain. 2018 Dec 1;141(12):3290-3307. doi: 10.1093/brain/awy281. PMID 30462175
- [Background] Mussigmann T, Bardel B, Lefaucheur JP. Resting-state electroencephalography (EEG) biomarkers of chronic neuropathic pain. A systematic review. Neuroimage. 2022 Sep;258:119351. doi: 10.1016/j.neuroimage.2022.119351. Epub 2022 Jun 2. PMID 35659993
- [Background] Ploner M, Sorg C, Gross J. Brain Rhythms of Pain. Trends Cogn Sci. 2017 Feb;21(2):100-110. doi: 10.1016/j.tics.2016.12.001. Epub 2016 Dec 23. PMID 28025007
- [Background] May ES, Nickel MM, Ta Dinh S, Tiemann L, Heitmann H, Voth I, Tolle TR, Gross J, Ploner M. Prefrontal gamma oscillations reflect ongoing pain intensity in chronic back pain patients. Hum Brain Mapp. 2019 Jan;40(1):293-305. doi: 10.1002/hbm.24373. Epub 2018 Sep 10. PMID 30260531
- [Background] Holsheimer J, Feenstra BW. Volume conduction and EEG measurements within the brain: a quantitative approach to the influence of electrical spread on the linear relationship of activity measured at different locations. Electroencephalogr Clin Neurophysiol. 1977 Jul;43(1):52-8. doi: 10.1016/0013-4694(77)90194-8. PMID 68872